CLINICAL TRIAL: NCT06210217
Title: Effect of Transesophageal Echocardiography-guided Non-fluid Limited Combined Dobutamine Strategy on Hepatic Venous Blood Flow Spectrum in Patients Undergoing Laparoscopic Hepatectomy: a Prospective Randomized Controlled Study
Brief Title: Effect of TEE-guided Non-fluid Limited Combined With Dobutamine on Hepatic Venous Blood Flow Spectrum
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Peng Liang，MD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023HX2017
Record Dates: First submitted 2024-01-04; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Laparoscopic Hepatectomy
MeSH Terms: interventions — Dobutamine; Injections; Saline Solution; Control Groups

STUDY DESIGN:
Intervention Model Description: In the dobutamine group, TEE will guide fluid rehydration to ensure preload, and dobutamine will be injected intravenously. In the control group, fluid will be limited by the principle of LCVP and the same amount of normal saline will be injected intravenously.
Who Masked: Participant, Outcomes Assessor
Masking Description: There are five groups (Participant, surgeon, anesthesiologist, data collector, outcome evaluator).
  Participants, surgeons, and outcome evaluators will be unaware of the grouping. Blinding will be maintained until data analysis is completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dobutamine group (Experimental): In the dobutamine group, 3~6μg/kg/min dobutamine will be injected intravenously after anesthesia induction until hemostasis is completed. To ensure preload, TEE will be used to monitor LVEDV and SV.
  Interventions: Drug: Dobutamine hydrochloride, Injectable
- Control group (Placebo Comparator): In the control group, 3mL/h normal saline will be injected intravenously after anesthesia induction until hemostasis is completed, and the liquid will be restricted according to the currently commonly used principle of LCVP, nitroglycerin can be used if necessary.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: Dobutamine hydrochloride, Injectable — In the dobutamine group, 3~6μg/kg/min dobutamine will be injected intravenously after anesthesia induction until hemostasis is completed. The dose of dobutamine will be increased if the operating field grade exceeds Grade II. Monitoring LVEDV and SV with TEE to ensure preload: after admission, the patient will be given 3-4 mL /kg/h equilibrium fluid as background infusion. LVEDV and SV will be monitored using TEE every 30 minutes after anesthesia induction. If LVEDV<75mL or SV<45mL, 200mL colloidal fluid will be given within 5min.
  Other Names: Dobutamine group
  Arms: Dobutamine group
Drug: 0.9% normal saline — In the control group, 3mL/h normal saline will be injected intravenously after anesthesia induction until hemostasis is completed. According to the currently commonly used principle of LCVP, the fluid will be limited to 3-4 ml /kg/h after anesthesia induction. If the operating field grade exceeds Grade II, nitroglycerin will be injected intravenously for remedial purposes at a rate of 0.3-0.8μg/kg/min.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Patients meeting enrollment criteria will be randomized 1:1 to either the dobutamine or the control group. In the dobutamine group, 3~6μg/kg/min dobutamine will be injected intravenously after anesthesia induction until hemostasis is completed. To ensure preload, transesophageal echocardiography (TEE) will be used to monitor left ventricular end-diastolic volume (LVEDV) and stroke volume (SV). In the control group, 3mL/h normal saline will be injected intravenously after anesthesia induction until hemostasis is completed, and the liquid will be restricted according to the currently commonly used principle of low central venous pressure(LCVP), nitroglycerin can be used if necessary.

DETAILED DESCRIPTION:
Patients meeting enrollment criteria will be randomized 1:1 to either the dobutamine or the control group.

Dobutamine group: 3~6μg/kg/min dobutamine will be injected intravenously after anesthesia induction until hemostasis is completed. The dose of dobutamine will be increased if the operating field grade exceeds Grade II. Monitoring LVEDV and SV with TEE to ensure preload: after admission, the patient will be given 3-4 mL /kg/h equilibrium fluid as background infusion. LVEDV and SV will be monitored using TEE every 30 minutes after anesthesia induction. If LVEDV<75mL or SV<45mL, 200mL colloidal fluid will be given within 5min.

Control group: 3mL/h normal saline will be injected intravenously after anesthesia induction until hemostasis is completed. According to the currently commonly used principle of LCVP, the fluid will be limited to 3-4 mL/kg/h after anesthesia induction. If the operating field grade exceeds Grade II, nitroglycerin will be injected intravenously for remedial purposes at a rate of 0.3-0.8μg/kg/min.

Dobutamine and nitroglycerin will be stopped after hemostasis, and the anesthesiologist will supplement the infusion according to his/her experience.

ELIGIBILITY:
Inclusion Criteria:

* undergo laparoscopic partial liver resection at West China Hospital from February 2024 to April 2024
* aged 18 to 65 years
* BMI<30kg/m2
* liver function Child-pugh grade A to B
* American Society of Anesthesiologists（ASA）grade Ⅰto Ⅲ.

Exclusion Criteria:

* coronary heart disease
* heart valvular disease
* arrhythmia
* stroke history
* cirrhosis
* esophageal varices
* esophageal disease, stomach disease, previous esophageal or gastric surgery history
* chronic kidney disease
* coagulation dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-07 (Estimated)

PRIMARY OUTCOMES:
Variation of hepatic venous blood flow spectrum | Intraoperative (after anesthesia induction, 10 minutes after the administration of dobutamine/normal saline, after pneumoperitoneum is established, and after hemostasis is completed.)
  The method of TEE monitoring hepatic vein blood flow: The TEE probe will be inserted into the patient's esophagus near the gastric fundus to show the liver. Next the probe will be rotated to the right to show the short axis of the inferior vena cava and the hepatic vein. Then the probe angle will be adjusted to 30-40° to show the long axis of the inferior vena cava and the hepatic vein, and the junction of the inferior vena cava and the hepatic vein. To record the blood flow spectrum of the hepatic vein using pulsed Doppler ultrasound (PW mode), the sampling volume should be placed in the hepatic vein, approximately 1.5-2cm away from the inferior vena cava opening. The angle between the sound beam and the blood flow direction should be less than 30°.
  The blood flow spectrum variation refers to the spectrum change measured at each time point relative to the basic spectrum after anesthesia induction.

SECONDARY OUTCOMES:
Intraoperative blood loss | intraoperative (Operation starts until hemostasis is completed.)
  Intraoperative blood loss can be calculated by adding the blood volume absorbed by gauze (8ml for small gauze, 25ml for medium gauze, and 50ml for large gauze) to the blood volume collected in the suction tank during the operation.
Surgical field grade | Intraoperative (When the liver parenchyma is transected after the pringle maneuver.)
  Grade Ⅰ is defined as the inferior vena cava and hepatic veins are very relaxed, and the liver section has little blood seepage, which is very easy to operate.
  Grade Ⅱ is defined as the inferior vena cava and hepatic vein are relaxed, and the liver section has less blood seepage, which is easy to operate.
  Grade Ⅲ is defined as the inferior vena cava and hepatic vein are tense, and the liver section oozes more blood, which is difficult to operate.
  Grade Ⅳ is defined as the inferior vena cava and hepatic vein are obviously tense, and the liver section oozes a lot of blood, which is very difficult to operate.
The remedy rate | Intraoperative (The liver parenchyma is transected until hemostasis is completed.)
  During hepatic parenchyma dissection, if the operating field grade is greater than grade II, the dobutamine dose (3-6 μg/kg/min) will be increased in the dobutamine group, and nitroglycerin (0.3-0.8μg /kg/min) will be added in the control group.
Duration of intraoperative hypotension | Intraoperative (From anesthesia induction to the patient leaving the operating room.)
  Intraoperative hypotension is defined as SBP<90mmHg, or MAP<60mmHg, or MAP/SBP decreasing greater than 20% of the baseline value during the perioperative period.
Ejection fraction | Intraoperative (anesthesia induction, 10 minutes after the administration of dobutamine/normal saline, after pneumoperitoneum is established, and after hemostasis is completed.)
  The ejection fraction will be measured by M-mode ultrasonography on the transgastric short-axis section of the left ventricle using TEE, recording the average value of three cardiac cycles.
The dose of vasoactive drugs | Intraoperative (From anesthesia induction to the patient leaving the operating room.)
  When perioperative SBP<90mmHg or MAP< 65mmHg, vasoactive drugs will be administered by the anesthesiologist.
Intraoperative urine volume | Intraoperative (anesthesia induction to the patient leaving the operating room.)
  After anesthesia induction, all patients will undergo catheterization to record urine volume during the operation.
Lactic acid | Intraoperative (after anesthesia induction, liver parenchyma transection is completed.)
  Invasive blood pressure will be monitored by the radial artery after anesthesia induction, and blood gas analysis will be performed after anesthesia induction and hepatic parenchyma dissection.
Length of operation | Intraoperative (From the beginning to the end of the surgery.)
  From the beginning to the end of the surgery.
Loss of hemoglobin | Preoperative and the third day after surgery.
  Preoperative hemoglobin content minus the hemoglobin content on the third day after surgery equals hemoglobin loss.
Loss of albumin | Preoperative and the third day after surgery.
  Preoperative albumin content minus the albumin content on the third day after surgery equals albumin loss.
Postoperative liver function (TB, ALT, AST) levels | The first and third day after surgery.
  The liver function (TB, ALT, AST) levels after surgery.
Incidence of AKI | Within 3 days after surgery
  AKI stage 1 is defined as serum creatinine(SCR) increases 1.5-2 times higher than the baseline.
  AKI stage 2 is defined as SCR is 2-3 times higher than the baseline.
  AKI stage 3 is defined as SCR increases by more than 3 times compared with the baseline.
Incidence of postoperative pulmonary complications | Up to 7days after surgery.
  Pulmonary complications include pulmonary infection, respiratory failure, and moderate or large pleural effusion.
Length of postoperative hospitalization | Up to 2 weeks after surgery.
  determined by the number of days from operation to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liang, Ph.D., Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No